CLINICAL TRIAL: NCT04236934
Title: Thoracentesis: Symptoms and Prediction of the Need for Therapeutic Thoracentesis: A Prospective Observational Study
Brief Title: Thoracentesis: Symptoms and Prediction of the Need for Therapeutic Thoracentesis
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 19-000067
Record Dates: First submitted 2019-12-19; First posted 2020-01-22 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pleural Effusion; Dyspnea; Patient Reported Outcomes; Diaphragm Movement; Ultrasound
MeSH Terms: conditions — Pleural Effusion; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All included patients: Patients with recurrent unilateral pleural effusion
  Interventions: Other: Assesment of diaphragm shape and diaphragm movement (by M-mode and the AREA-method) by ultrasound before and after thoracentesis

INTERVENTIONS:
Other: Assesment of diaphragm shape and diaphragm movement (by M-mode and the AREA-method) by ultrasound before and after thoracentesis — Questionnaire is about symptoms measured by Edmonton Symptom Assessment Score (ESAS) and dyspnea also by modified Borg Scale (MBS)
  Other Names: A questionnaire before and after thoracentesis and daily until next therapeutic thoracentesis

SUMMARY:
Recurrent fluid surrounding the lungs is associated with poor quality of life, the main symptom being dyspnea. These patients are in need of recurrent removal of the fluid using drainage. The mechanism causing dyspnea is not fully understood.

By using ultrasound to evaluate the movement of the diaphragm before and after removal of fluid and the patients symptoms before removal of fluid and until next removal the research group aims to clarify the temporal development in symptoms and the role of the diaphragm.

The researchers will also evaluate the ability of the pulmonologist and patient to predict when the patient will need the next removal of fluid in patients with recurrent unilateral pleural effusion.

DETAILED DESCRIPTION:
Recurrent pleural effusion (PE) is associated with impaired quality of life, the main symptom being dyspnea. The mechanisms causing dyspnea in PE is not fully understood. These patients are in need of recurrent therapeutic thoracentesis.

By evaluating the movement of diaphragma before and after thoracentesis and measure the patients symptoms before thoracentesis and until the next thoracentesis the researchers aim to clarify the temporal development in symptoms and the role of the diaphragm.

The researchers will also evaluate the ability of the pulmonologist and patient to predict when the patient will need the next therapeutic thoracentesis in patients with recurrent unilateral pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Unilateral pleural effusion.
* A minimum of two thoracentesis prior to inclusion.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Bilateral pleural effusions.
* Inability to understand written or spoken Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Pleura Clinic (an outpatient clinic in the Department of Pulmonary Disease) at Næstved Sygehus or Zealand University Hospital, Roskilde (the two regional centers for work up of pulmonary malignancy). Patients are referred from the general practitioner or from other hospital departments both Næstved Sygehus and other hospitals.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Difference between time to next thoracentesis scheduled by the pulmonologist and patient respectively versus time to patient-reported need for thoracentesis | At the day of the next thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  Measured in days. The patients and pulmonologists scheduling is recorded on a questionnaire at the day of first thoracentesis, after the procedure

SECONDARY OUTCOMES:
Patients experienced well being | At day 1 immediately prior to and immediately after thoracentesis
  Symptoms measured by ESAS (Edmonton Symptom Assessment System, contains visual analogue scales measuring tiredness, pain, drowsiness, nausea, appetite, dyspnea, depression, anxiety, and general well being, scale 0-10, 0 being no symptoms, 10 being the worse symptoms)
Patients perception of dyspnea | At day 1 immediately prior to and immediately after thoracentesis.
  Symptoms measured by MBS (Modified Borg Scale, scale1-5, 1 being no dyspnea, 5 being the worse dyspnea)
Patients perception of dyspnea | At day 1 immediately prior to and immediately after thoracentesis.
  Symptoms measured by MRC (Medical Research Council Dyspnoea Scale, scale1-5, 1 being the least dyspnea, 5 being the worse dyspnea)
Patient experienced dyspnea until next thoracentesis | At the day of the next thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  Measured in a daily diary completed at the same time slot every day by MBS (Modified Borg Scale, scale1-5, 1 being no dyspnea, 5 being the worse dyspnea)
Patient experienced dyspnea until next thoracentesis | At the day of the next thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  Measured in a daily diary completed at the same time slot every day by Measured in a daily diary completed at the same time slot every day by MRC (Medical Research Council Dyspnoea Scale, scale1-5, 1 being the least dyspnea, 5 being the worse dyspnea)
Patient experienced well being until next thoracentesis | At the day of the next thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  Measured in a daily diary completed at the same time slot every day by ESAS Symptoms measured by ESAS (Edmonton Symptom Assessment System, contains visual analogue scales measuring tiredness, pain, drowsiness, nausea, appetite, dyspnea, depression, anxiety, and general well being, scale 0-10, 0 being no symptoms, 10 being the worse symptoms)
Fluid removed at the first study-thoracentesis | At day 1, immediately after end of procedure
  measured in mL.
Fluid removed at the second study-thoracentesis | At the day of the the second thoracentesis, immediately after end procedure
  measured in mL.
Correlation between amount of pleural fluid removed at the first study-thoracentesis (outcome 6) and symptoms (well being and dyspnea, outcome 4 and 5) until next thoracentesis. | At the day of the next thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  amount of fluid measured in mL.
Correlation between patient's symptoms (well being and dyspnea, outcome 4, 5and 6) and time to next thoracentesis | At the day of the next thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  Time measured in days
Correlation between time in between thoracentesis and amount of fluid drained at the following thoracentesis | thoracentesis or 2 months after the first study-thoracentesis, whichever comes first.
  Time measured in days and amount of fluid measured in mL
Correlation between well being and dyspnea (outcome 2, 3 and 4) and findings on lung ultrasound before and after completed thoracentesis | At day 1 immediately after ended procedure
  Diaphragmatic movement (measured by M-mode and "The Area method", diaphragmatic shape (convex, flat, concave) and Septae-score)

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Bødtger, MD, PhD, Principal Investigator — Department of Pulmonary Medicin, Næstved Sygehus
Locations (2):
- Denmark (2):
  - Næstved Sygehus, department of pulmonary medicine, Næstved, Region Sjælland
  - Zealand University Hospital, Roskilde, Roskilde, Region Sjælland